CLINICAL TRIAL: NCT02647892
Title: Optimal Lidocaine Buffering to Reduce Injection Pain in Local Anesthesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB protocol administratively closed, Continuing Review or Study Completion Report not submitted
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0787-15-EP
Record Dates: First submitted 2015-12-17; First posted 2016-01-06 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Local Anesthesia
MeSH Terms: interventions — Lidocaine; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Active Comparator): 10 mg/mL lidocaine; Frequency: 1
  Interventions: Drug: lidocaine
- Arm B (Active Comparator): 9 mg/mL of 10% sodium bicarbonate-90% lidocaine; Frequency: 1
  Interventions: Drug: lidocaine; Drug: sodium bicarbonate
- Arm C (Active Comparator): 7.5 mg/Ml of 25% sodium bicarbonate-75% lidocaine Frequency: 1
  Interventions: Drug: lidocaine; Drug: sodium bicarbonate
- Arm D (Active Comparator): 5 mg/mL 50% sodium bicarbonate-50% lidocaine Frequency: 1
  Interventions: Drug: lidocaine; Drug: sodium bicarbonate

INTERVENTIONS:
Drug: lidocaine — local anesthesia
  Other Names: xylocaine
Drug: sodium bicarbonate — additional drug added to lidocaine
  Arms: Arm B; Arm C; Arm D

SUMMARY:
The purpose of this study is to determine the optimal amount of lidocaine buffering needed to decrease injection pain when administering local anesthesia.

DETAILED DESCRIPTION:
Once the site is chosen, the skin will be anesthetized as usual. This study will utilize a commercially prepared 1% lidocaine solution mixed with standard sodium bicarbonate. A total of 10 mL will be used.

ELIGIBILITY:
Inclusion Criteria:

* adults presenting for routine thyroid biopsy, paracentesis or thoracentesis in interventional radiology

Exclusion Criteria:

* Patients requiring sedation
* Patients with altered mental status
* Children
* Patients allergic to lidocaine or sodium bicarbonate

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Injection pain | 6 months
  numeric pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McBride, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skarsvag TI, Wago KJ, Tangen LF, Lundbom JS, Hjelseng T, Ballo S, Finsen V. Does adjusting the pH of lidocaine reduce pain during injection? J Plast Surg Hand Surg. 2015 Oct;49(5):265-267. doi: 10.3109/2000656X.2015.1047780. Epub 2015 May 19. PMID 25991379
- [Background] Bartfield JM, Gennis P, Barbera J, Breuer B, Gallagher EJ. Buffered versus plain lidocaine as a local anesthetic for simple laceration repair. Ann Emerg Med. 1990 Dec;19(12):1387-9. doi: 10.1016/s0196-0644(05)82603-4. PMID 2240750
- [Background] Colaric KB, Overton DT, Moore K. Pain reduction in lidocaine administration through buffering and warming. Am J Emerg Med. 1998 Jul;16(4):353-6. doi: 10.1016/s0735-6757(98)90126-7. PMID 9672449
- [Background] Orlinsky M, Hudson C, Chan L, Deslauriers R. Pain comparison of unbuffered versus buffered lidocaine in local wound infiltration. J Emerg Med. 1992 Jul-Aug;10(4):411-5. doi: 10.1016/0736-4679(92)90269-y. PMID 1430977
- [Background] Matsumoto AH, Reifsnyder AC, Hartwell GD, Angle JF, Selby JB Jr, Tegtmeyer CJ. Reducing the discomfort of lidocaine administration through pH buffering. J Vasc Interv Radiol. 1994 Jan-Feb;5(1):171-5. doi: 10.1016/s1051-0443(94)71478-0. PMID 8136599
- [Background] Machin D, Campbell M, Fayers P, Pinol A. 1997. Sample Size Tables for Clinical Studies, 2nd Edition. Blackwell Science. Malden MA.